CLINICAL TRIAL: NCT03281707
Title: Evaluation of NIRS and DO2i Correlation and Their Relationship With Organ Failure During Cardiac Surgery: a Prospective Monocentric Study.
Brief Title: NIRS and DO2i Correlation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Principal Investigator, luca salvi, Anesthesia and ICU director, Centro Cardiologico Monzino
Other Study IDs: R627/17-CCM 662
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Multiorgan Failure; Perfusion; Complications
Keywords: NIRS; DO2
MeSH Terms: conditions — Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: NIRS — NIRS devices patch will be applied on patients' head in order to measure the cerebral saturation of each cerebral emisphere
Other: DO2i — Oxygen delivery standardized to the body surface area will be calculate in order to optimize tissue perfusion

SUMMARY:
This study evaluates the association between near infrared spectroscopy (NIRS) and indexed oxygen delivery (DO2i) and their possible correlation with postoperative organ failure.

DETAILED DESCRIPTION:
Literature evidences show that levels of DO2i under 262-272 mL/min/m2 during cardiopulmonary by-pass (CPB) are associated with an increased incidence of acute kidney injury (AKI).

Furthermore, it has been demonstrated that keeping a NIRS of 75-80% compared to the basal value reduces the risk of perioperative morbidity. On the other hand, a NIRS < 50% of basal value seems to be predictive of an increase in morbidity.

All of those studies had been performed during CPB and knowledge lacks in management of DO2i and NIRS before and after CPB.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing cardiac surgery with cardiopulmonary by-pass whose have been signed the consent informed

Exclusion Criteria:

* Impossibilty to collect a correct continuous cardiac output measure with PiCCO (chronic atrial fibrillation or severe peripheral vasculopaty)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-09-30 (Estimated); Primary Completion 2018-10-30 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the correlation between NIRS and DO2i during cardiac surgery | Intraoperative

SECONDARY OUTCOMES:
Evaluate the correlation between NIRS, DO2i and SOFA score | 7 days postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Luca Salvi, MD, Principal Investigator — Centro Cardiologico Monzino

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ranucci M, Romitti F, Isgro G, Cotza M, Brozzi S, Boncilli A, Ditta A. Oxygen delivery during cardiopulmonary bypass and acute renal failure after coronary operations. Ann Thorac Surg. 2005 Dec;80(6):2213-20. doi: 10.1016/j.athoracsur.2005.05.069. PMID 16305874
- [Result] de Somer F, Mulholland JW, Bryan MR, Aloisio T, Van Nooten GJ, Ranucci M. O2 delivery and CO2 production during cardiopulmonary bypass as determinants of acute kidney injury: time for a goal-directed perfusion management? Crit Care. 2011 Aug 10;15(4):R192. doi: 10.1186/cc10349. PMID 21831302
- [Result] Nielsen HB, Borglum J. Cerebral oxygenation in heart surgery. Anesth Analg. 2007 Aug;105(2):537; author reply 538-9. doi: 10.1213/01.ane.0000265698.02800.d4. No abstract available. PMID 17646526
- [Result] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239